CLINICAL TRIAL: NCT02451709
Title: Can Electronic Adherence Monitors With Feedback and Daily Reminders Improve Adherence and Health Outcomes in Children With Asthma?
Brief Title: STudy of Asthma Adherence Reminders
Acronym: STAAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SCH/13/041
Record Dates: First submitted 2015-05-05; First posted 2015-05-22 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-05

CONDITIONS: Childhood Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feedback and alarms (Experimental): Standard education about importance of inhaled steroids and regular adherence to inhaled steroids after recruitment to study.
  Randomized to receive an electronic adherence device ( activated smartinhaler or smartturbo - Nexus 6) with twice daily alarm reminders activated. Patient decides times, different times on weekdays and weekends if required. This device fitted to their regular preventer inhaler, patient aware of its presence and its purpose in the context of the study.
  Reviewed in standard asthma clinic every 3 months for 12 months. At each clinic visit, adherence information downloaded from device and data shared with patient and family (feedback of adherence data). Discussion about adherence rates, and action planning for the next 3 months to improve adherence if necessary.
  Interventions: Device: Activated Smartinhaler or Smartturbo; Other: Feedback of adherence data
- No feedback or alarms (Active Comparator): Standard education about importance of inhaled steroids and regular adherence to inhaled steroids after recruitment to study.
  Randomized to receive an electronic adherence device. Deactivated Smartinhaler or Smartturbo.
  Device not activated to play reminder alarms. This device fitted to their regular preventer inhaler, patient aware of its presence and its purpose in the context of the study.
  Reviewed in standard asthma clinic every 3 months for 12 months. At each clinic visit, adherence information downloaded from device but data not shared with patient, and no adherence discussion.
  Interventions: Device: Deactivated Smartinhaler or Smartturbo

INTERVENTIONS:
Device: Activated Smartinhaler or Smartturbo — Medication reminder alarms
  Other Names: Electronic adherence monitor
  Arms: Feedback and alarms
Other: Feedback of adherence data — Review of adherence data with action planning
  Arms: Feedback and alarms
Device: Deactivated Smartinhaler or Smartturbo — Alarms deactivated and no feedback
  Other Names: Electronic adherence monitor
  Arms: No feedback or alarms

SUMMARY:
To determine whether electronic adherence monitoring with feedback and reminder alarms can improve adherence and health outcomes in childhood asthma.

DETAILED DESCRIPTION:
This study will investigate whether adding an electronic adherence monitor to inhaled steroids, and feeding this information back to patients and families can improve adherence and outcomes in childhood asthma. The devices will also sound twice daily reminder alarms to act as direct medication prompts. This intervention will be compared to a control group in which adherence is monitored, but with no feedback or alarms.

ELIGIBILITY:
Inclusion Criteria:

* Doctor diagnosed asthma.
* On at least BTS stage 2, which means they will be on regular inhaled steroids.
* No change in regular asthma treatment in the last 1 month (on regular inhaled steroids, no change in steroid dose for

  1 month, no change in add on therapy in the last month).
* ACQ (Asthma Control Questionnaire) score more than or equal to 1.5.
* Can speak and understand English.

Exclusion Criteria:

* BTS stage 5 asthma (complex issues, too unstable).
* Recent changes to asthma treatment within the last month. (see above)
* ACQ (Asthma Control Questionnaire) score < 1.5.
* Another chronic health condition (eg diabetes, congenital heart disease, cystic fibrosis).
* Can't speak or understand English.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in asthma control from baseline at 3 months | 3 months
  Recorded as an Asthma Control Questionnaire (ACQ) score.Mean score of 0 -7, lower score indicating better asthma control.
Change in asthma control from baseline at 6 months | 6 months
  Recorded as an Asthma Control Questionnaire (ACQ) score.Mean score of 0 -7, lower score indicating better asthma control.
Change in asthma control from baseline at 9 months | 9 months
  Recorded as an Asthma Control Questionnaire (ACQ) score.Mean score of 0 -7, lower score indicating better asthma control.
Change in asthma control from baseline at 12 months | 12 months
  Recorded as an Asthma Control Questionnaire (ACQ) score.Mean score of 0 -7, lower score indicating better asthma control.

SECONDARY OUTCOMES:
Asthma-related quality of life, as measured by the "Mini Paediatric Asthma Quality of Life Questionnaire" (Mini PAQLQ) | Recorded at baseline, 3, 6, 9 and 12 months.
  Mean score of 0-7, lower score indicating poorer asthma - related quality of life.
Parents' illness perceptions as measured by the "brief illness perception questionnaire. | Recorded at baseline
  As measured by the "brief illness perception questionnaire. A higher score indicates a more threatening view of the illness.
Unplanned GP/ ED attendances for asthma | Recorded at baseline, 3, 6, 9 and 12 months.
  Number of unplanned visits to GP or A&E for asthma in the previous 3 months.
Rescue beta-agonist use | Recorded at baseline, 3, 6, 9 and 12 months.
  Question score on the ACQ regarding recent beta agonist use.
Adherence to ICS treatment | Recorded at baseline, 3, 6, 9 and 12 months.
  Electronic adherence rate as measured by the smartinhaler or smartturbo. Adherence rate calculated as percentage of prescribed doses actually taken. Adherence rate capped at 100% for any single day.
Level of maintenance asthma therapy. Treatment level (modified BTS step) at 12 months and individual change in modified BTS step between baseline and 12 months | Recorded at baseline, 3, 6, 9 and 12 months.
  Dose of ICS
Forced Expiratory Volume in 1 second (FEV1) - % predicted | Recorded at baseline, 3, 6, 9 and 12 months.
  % predicted value compared with Global Lung Initiative 2012 reference values.
Medication beliefs | Recorded at baseline
  As measured by the "beliefs about medicines" questionnaire. A higher score indicates multiple concerns and doubts about inhaled steroids.
Rescue doses of oral steroids | Recorded at baseline, 3, 6, 9 and 12 months.
  Number of rescue doses of oral steroids required in the previous 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Morton, Principal Investigator — Investigator
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, Sheffield (South Yorkshire District), United Kingdom

REFERENCES:
- [Derived] Morton RW, Elphick HE, Rigby AS, Daw WJ, King DA, Smith LJ, Everard ML. STAAR: a randomised controlled trial of electronic adherence monitoring with reminder alarms and feedback to improve clinical outcomes for children with asthma. Thorax. 2017 Apr;72(4):347-354. doi: 10.1136/thoraxjnl-2015-208171. Epub 2016 Nov 4. PMID 27815524